CLINICAL TRIAL: NCT02811354
Title: Phase II Study of AZD9291 in Patients With Advanced Stage Non-small Cell Lung Cancer Following Prior EGFR TKI Therapy With EGFR and T790M Mutations Detected in Plasma Circulating Tumor DNA (PLASMA)
Brief Title: Phase II Study of AZD9291 in Advanced Stage NSCLC With EGFR and T790M Mutations Detected in Plasma Ct-DNA
Acronym: PLASMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: AstraZeneca (Industry); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-10932; 2015/01069 (Other: NHG DSRB)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD9291 (Experimental): Patient will be treated with AZD9291 at a starting dose of 80mg once a day until the patient completes the study, withdraws from the study or closure of the study. A cycle of treatment is defined as 28 days of once daily AZD9291 treatment. Patients may continue to receive AZD9291 until objective disease progression (determined by RECIST 1.1) or if the subject is no longer receiving clinical benefit in the Investigator's opinion.
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — oral administration as a single daily dose of 80 mg
  Other Names: Osimertinib

SUMMARY:
Circulating tumor DNA (ctDNA) is a highly specific and effective biomarker for the detection of EGFR mutation status. We hypothesise AZD9291 is efficacious in patients with EGFR sensitizing mutations and T790M detected in plasma ctDNA.

This is a prospective, open label, multi-centre single arm phase II study assessing the efficacy and safety of AZD9291 monotherapy in patients with stage IIIB or IV harboring sensitising EGFR mutation (exon 19 deletions or exon 21 L858R substitution mutations) and T790M who have progressed following prior treatment with an approved EGFR TKI. Approximately 106 subjects will be enrolled.

All patients must have documented radiological progression on EGFR-TKI treatment and on the last treatment administered prior to enrolling in the study.

DETAILED DESCRIPTION:
As T790M is the most common mechanism of acquired resistance to EGFR TKI, EGFR TKIs targeting T790M has been developed.

AZD9291 is an oral, potent, irreversible EGFR-TKI selective for sensitizing (EGFRm) and T790M resistance mutation with a significant selectivity margin against wild-type EGFR. As a result, AZD9291 can effectively block EGFR signaling both in EGFR single mutant cells with activating EGFR mutations and in double mutant cells bearing the resistance T790M mutation.

This is a prospective, open label, multi-centre single arm phase II study assessing the efficacy and safety of AZD9291 monotherapy in patients with stage IIIB or IV harboring sensitising EGFR mutation (exon 19 deletions and exon 21 L858R substitution mutations) and T790M who have progressed following prior treatment with an approved EGFR TKI. Approximately 108 subjects will be enrolled.

All patients must have documented radiological progression on EGFR-TKI treatment and on the last treatment administered prior to enrolling in the study.

Target patient population:

Patients will be > 18 years of age, with a diagnosis of locally advanced/metastatic NSCLC not amenable to curative surgery or radiotherapy with documented activating EGFR mutations (exon 19 deletions and exon 21 L858R substitution mutations) at the time of initial diagnosis, have radiological disease progression following either 1st line EGFR TKI treatment OR following prior therapy with an EGFR TKI and a platinum-based doublet chemotherapy. Plasma sample must harbour an EGFR mutation known to be associated with EGFR TKI sensitivity (exon 19 deletion, L858R as well as presence of T790M by central lab testing from a plasma sample taken after confirmation of disease progression on the most recent treatment regimen. Patients must have normal organ and bone marrow function and ECOG PS 0-2.

Treatment and regimens:

Patient will be treated with AZD9291 at a starting dose of 80mg once a day until the patient completes the study, withdraws from the study or closure of the study. A cycle of treatment is defined as 28 days of once daily AZD9291 treatment. Patients may continue to receive AZD9291 until objective disease progression (determined by RECIST 1.1) or if the subject is no longer receiving clinical benefit in the Investigator's opinion.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients must be >= 21 years of age.
3. Locally advanced/metastatic NSCLC not amenable to curative surgery or radiotherapy
4. Documentation of activating EGFR mutations (exon 19 deletions or exon 21 L858R substitution mutations) at the time of initial diagnosis
5. Radiological documentation of disease progression: following 1st line EGFR TKI treatment but who have not received further treatment OR following prior therapy with an EGFR TKI and a platinum-based doublet chemotherapy. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
6. Patient may receive up to two lines of therapies (including EGFR TKI).
7. Plasma sample must harbour an EGFR mutation known to be associated with EGFR TKI sensitivity (exon 19 deletion, L858R). Confirmation of T790M status by central lab testing from a plasma sample taken after confirmation of disease progression on the most recent treatment regimen.
8. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin >= 10.0 g/dL and no blood transfusions in the 28 days prior to entry
   * Absolute neutrophil count (ANC) >= 1.5 x 109/L
   * No features suggestive of MDS/AML on peripheral blood smear
   * White blood cells (WBC) > 3x109/L
   * Platelet count >= 100 x 109/L
   * Total bilirubin <= 1.5 x institutional upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) <= 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be <= 5x ULN
   * Serum creatinine <= 1.5 x institutional upper limit of normal (ULN)
   * ECOG performance status 0-2
9. Patients must have a life expectancy >= 12 weeks.
10. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
11. Male patients should be willing to use barrier contraception (see Restrictions, Section 5.1)
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
13. At least one lesion, not previously irradiated, that can be accurately measured at baseline as >= 10 mm in the longest diameter (except lymph nodes which must have short axis >= 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Treatment with an EGFR-TKI within 8 days of study entry; any cytotoxic chemotherapy, or other anticancer drugs within 21 days of study entry
3. Treatment with an investigational drug within five half-lives of the compound
4. Prior treatment with an immune checkpoint inhibitor
5. Previous treatment with AZD9291 (or 3rd generation EGFR TKIs)
6. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for >= 5 years
7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks
8. The patient may receive bisphosphonates for the treatment of bone metastases.
9. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
10. Unstable spinal cord compression/brain metastases unless asymptomatic, stable and not requiring steroids for at least 2 weeks prior to start of study treatment.
11. Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
12. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior) (Appendix A). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
13. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
14. Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
15. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
16. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9291
17. History of hypersensitivity to AZD9291 (or drugs with a similar chemical structure or class to AZD9291) or any excipients of these agents
18. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive serum pregnancy test prior to study entry
19. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
20. Previous allogeneic bone marrow transplant.
21. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-02-24 (Estimated); Study Completion 2020-02-24 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the time of their first treatment with daily AZD9291 till 28 days after discontinuation

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the time of their first treatment with daily AZD9291 till 28 days after discontinuation
Duration of response (DoR) | From the time of their first treatment with daily AZD9291 till 28 days after discontinuation
Disease control rate (DCR) | From the time of their first treatment with daily AZD9291 till 28 days after discontinuation
Tumour shrinkage | From the time of their first treatment with daily AZD9291 till 28 days after discontinuation
Overall survival (OS) | From the time of their first treatment with daily AZD9291 till 28 days after discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Ross Soo, Principal Investigator — National University Hospital, Singapore
Locations (8):
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Prince of Wales Hospital, Shatin
- National University Hospital, Singapore, Singapore
- South Korea (3):
  - Samsung Medical Center Sungkyunkwan University, Irwon-dong, Seoul
  - Yonsei Cancer Center, Sinchon-dong, Seoul
  - Seoul National University College of Medicine, Yeongeon-dong, Seoul
- National Taiwan University Hospital, Taipei, Taiwan
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang T, Zhou C. Clinical activity of the mutant-selective EGFR inhibitor AZD9291 in patients with EGFR inhibitor-resistant non-small cell lung cancer. Transl Lung Cancer Res. 2014 Dec;3(6):370-2. doi: 10.3978/j.issn.2218-6751.2014.08.02. PMID 25806323
- [Background] Cross DA, Ashton SE, Ghiorghiu S, Eberlein C, Nebhan CA, Spitzler PJ, Orme JP, Finlay MR, Ward RA, Mellor MJ, Hughes G, Rahi A, Jacobs VN, Red Brewer M, Ichihara E, Sun J, Jin H, Ballard P, Al-Kadhimi K, Rowlinson R, Klinowska T, Richmond GH, Cantarini M, Kim DW, Ranson MR, Pao W. AZD9291, an irreversible EGFR TKI, overcomes T790M-mediated resistance to EGFR inhibitors in lung cancer. Cancer Discov. 2014 Sep;4(9):1046-61. doi: 10.1158/2159-8290.CD-14-0337. Epub 2014 Jun 3. PMID 24893891